CLINICAL TRIAL: NCT03370224
Title: Application of the Modified Story Memory Technique (mSMT)© to Aging
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director, Neuropsychology and Neuroscience Research, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-990-17
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Aging; Mild Cognitive Impairment
Keywords: Memory; Learning; Cognition; Treatment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive memory retraining exercises administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Memory retraining exercises
- Placebo (Placebo Comparator): The placebo group will receive placebo control memory exercises administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Interventions: Behavioral: Placebo control memory exercises

INTERVENTIONS:
Behavioral: Memory retraining exercises — Memory retraining exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: Experimental Group
Behavioral: Placebo control memory exercises — Placebo control memory exercises will be administered on a laptop computer twice a week for 5 weeks (10 training sessions).
  Arms: Placebo

SUMMARY:
This study is a double-blind placebo-controlled randomized clinical trial (RCT) to provide Class I evidence in support of or in refute of the efficacy of the modified Story Memory Technique (mSMT) in healthy aging (HA)and in persons with mild cognitive impairment (MCI). Outcomes will be measured through three mechanisms: (1) a traditional neuropsychological evaluation (NPE) (2) an assessment of global functioning (AGF) examining the impact of the treatment on daily activities, and (3) an optional functional magnetic resonance imaging (fMRI) scan.

DETAILED DESCRIPTION:
Studies conducted at Kessler Foundation (KF) have demonstrated the modified Story Memory Technique (mSMT) to be effective for improving new learning in individuals with MS and TBI. Efficacy of the individualized mSMT has been clearly demonstrated across three realms of functioning, objective behavior, brain functioning and everyday life in multiple RCTs with both MS and TBI samples. This convincing data provides Class I evidence supporting the efficacy of the individual mSMT for improving new learning and memory in MS with documentation of long-lasting treatment effects on both standardized learning tests and neuroimaging. Current work with the mSMT is focusing on a group administration format, with a RCT funded by the Department of Defense.

Ongoing work in healthy aging (HA), led by George Rebok, PhD at the Johns Hopkins School of Public Health, has applied cognitive retraining to older healthy adults. Multiple, strong rationale for pursuing such applications of cognitive rehabilitation include the fact that the 65 and older population is growing (an estimated 20% of population (72 million) will be 65 and older by 2030), cognitive decline is most feared aspect of growing older, drug trial results addressing this challenge have been disappointing and, most importantly, cognitive impairments heavily affect the aging population. Specifically, 1 in 4 adults 70 years or older have a cognitive impairment without dementia and roughly 5.3 million people in the U.S. have Alzheimer's disease. Rebok and colleagues have applied Speed of Processing Training to a large cohort of healthy older adults (age 65+) and found a 33-48% risk reduction of dementia onset 10 years post treatment. These encouraging results suggest that providing cognitively enhancing treatments prior to the onset of dementia may in fact stave off the dementia process and provide older individuals with more years free of cognitive deficit.

Given the substantial success of the mSMT in improving new learning and memory functioning in persons with TBI and MS, we seek to apply the mSMT to an aging population with multiple aims.

Aim 1. Examine the efficacy of the mSMT to increase learning and memory abilities in older adults with mild cognitive impairment (MCI) and older adults with no signs of cognitive impairment (healthy aging group: HA).

Aim 2. Examine the long term impact of the mSMT on new learning and memory abilities one and two years post-intervention for both the MCI group and the HA group.

Aim 3. Examine the impact of early cognitive enhancement with the mSMT on measures of daily life functioning and overall quality of life immediately posttreatment and at each follow-up assessment.

Aim 4. Examine the neural correlates during encoding and retrieval associated with early cognitive enhancement from the mSMT immediately post-treatment and at each follow-up assessment

To achieve these goals, we will recruit 40 individuals over the age of 65 to participate in the study. Each participant will undergo baseline cognitive assessment. Based on the assessment results, he / she will be allocated to the HA block or the MCI block. Within each block, participants will be randomized to a treatment group or a placebo control group. The treatment group will undergo 10 sessions of the mSMT, while the placebo control group will undergo 10 sessions of memory exercises. We have used this placebo condition in multiple randomized clinical trials in the past, with success. Repeat assessments will then occur within one week of completing treatment, 6 months after completing treatment, one year after completing treatment, 2 years after completing treatment and 6 years after treatment. Each assessment will evaluate new learning and memory abilities as well as multiple other aspects of cognitive functioning through a neuropsychological assessment (NP). Participants will also complete an assessment of global functioning (AGF) which evaluates cognitive functioning in daily life. In addition, we will collect neuroimaging data on a subsample of participants willing and able to complete imaging procedures

ELIGIBILITY:
Inclusion Criteria:

* older than 65
* primary language is English.

Exclusion Criteria:

* diagnosis of any neurological condition (Alzheimer's disease, dementia, stroke, multiple sclerosis, Brain Injury, Parkinson's disease, etc.).
* diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder.
* abuse of illicit drug within the past 6 months.

For optional MRI

* pacemaker or other implanted electrical device, brain stimulator, aneurysm clip (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids [cochlear implants]), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* dental implants
* left handed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in scores on standardized neuropsychological tests of memory using the California Verbal Learning Test | Scores will be assessed at five time-points: Baseline (week 1), immediately post-intervention (week 7) and 6, 12, 24 months, and 6 years post-intervention.
  California Verbal Learning Test

SECONDARY OUTCOMES:
Change in scores on self-report of emotional functioning, measured via the Chicago multiscale depression inventory | Scores will be assessed at five time-points: Baseline (week 1), immediately post-intervention (week 7) and 6, 12 ,24 months and 6 years post-intervention]
  Chicago multiscale depression inventory
Change in scores on self-report of memory functioning, measured via questionnaire by the Memory Functioning Questionnaire | Scores will be assessed at five time-points: Baseline (week 1), immediately post-intervention (week 7) and 6, 12, 24 months and 6 years post-intervention]
  Memory Functioning Questionnaire
Change in scores on self-report of quality of life, measured via the SF-12 | Scores will be assessed at five time-points: Baseline (week 1), immediately post-intervention (week 7) and 6, 12 and 24 months and 6 years post-intervention]
  SF -12

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No